CLINICAL TRIAL: NCT06697522
Title: A Randomized, Double-masked, Placebo-controlled, Parallel-group Study of Safety and Efficacy of Atropine Sulfate Eye Drops (0.01%) in the Treatment of Near-work-induced Transient Myopia (NITM) in Children
Brief Title: Study of Atropine Sulfate Eye Drops(0.01%) in Treating Near-work-induced Transient Myopia in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ocumension Therapeutics (Suzhou) Co., Ltd (Industry)
Collaborators: Beijing Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Protocol V 7.0
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Myopia
Keywords: Atropine
MeSH Terms: conditions — Myopia | interventions — Atropine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.01% Atropine (Experimental): Atropine Sulfate Eye Drops, conc. 0.01%
  Interventions: Drug: Atropine Sulfate
- Blank Solvent (Placebo Comparator): Blank solvent placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atropine Sulfate — low concentration atropine (0.01%)
  Other Names: Investigational product
  Arms: 0.01% Atropine
Drug: Placebo — Blank comparator
  Other Names: Blank Solvent
  Arms: Blank Solvent

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, parallel-group study to evaluate the safety and efficacy of atropine sulfate eye drops (0.01%) in treating transient myopia induced by near work tasks (NITM) in pediatric subjects.

DETAILED DESCRIPTION:
All eligible subjects will be randomly assigned in a 1:1 ratio to either the 0.01% atropine sulfate eye drops group or the atropine sulfate eye drops vehicle placebo control group. Subjects in the treatment group will apply one drop of 0.01% atropine sulfate eye drops to each eye before going to bed at night, while subjects in the control group will apply one drop of the atropine sulfate eye drops vehicle placebo to each eye before going to bed at night. All eligible subjects will be randomly grouped and receive treatment for a period of 12 weeks. All subjects will be followed up according to the same timing and examination schedule. The follow-up time points will be on the 1st day, 14th day, and 12th week after administration, as well as 12 weeks after discontinuation of the medication.

ELIGIBILITY:
Inclusion Criteria:

1. For subjects of age between 6 to 8, their parents or legal guardians must provide written informed consent; For 8 year old subjects and above, both the subjects and their legal guardians need to sign the informed consent form.
2. They must be able to comply with the research requirements, attend all study visits, and be accompanied by their parents/legal guardians.
3. The age range during the screening period (from Day -14 to Day 0) is 6-15 years, with no gender restrictions.
4. The optometry results during the screening period should show: a) Myopia between -0.50DS and -4.00DS. b) Astigmatism ≤1.50DC, and less than half of the spherical lens power. c) The initial NITM value (equivalent sphere) for either eye should be ≤-0.40D.
5. The difference in refractive error between both eyes during the screening period should be ≤1.00D in equivalent spherical lens power.
6. The best corrected visual acuity (BCVA) for both eyes during the screening period should be ≥0.8 on the standard logarithmic visual acuity chart.
7. They must be able and willing to avoid using all prohibited medications during the washout period between screening and randomization, as well as during the study period, with no significant risk to the subjects.

Exclusion Criteria:

1. Known contraindications or allergies to atropine sulfate, the study drug, or its components.
2. Clinically significant abnormal findings on slit-lamp microscopy examination (e.g., cataract) that may affect the measurement of best-corrected visual acuity in either eye at the time of screening, or known clinically significant findings from a previous slit-lamp microscopy examination in either eye.
3. Clinically significant abnormal findings on direct ophthalmoscopy at the time of screening in either eye, or known previous clinically significant retinal findings in either eye.
4. Evidence of any ocular motility disorder or restriction of extraocular muscle movement (e.g., nystagmus).
5. Presence of infectious eye diseases (such as bacterial, viral, or fungal infections).
6. Active ocular inflammation in either eye or a history of chronic or recurrent ocular inflammation (e.g., moderate to severe blepharitis, allergic conjunctivitis, peripheral ulcerative keratitis).
7. History of ocular herpes virus infection, iritis, scleritis, or uveitis, regardless of whether it is active at the time of screening.
8. Abnormal pupillary light reflex and/or amblyopia at the time of screening.
9. Intraocular pressure (IOP) in either eye <9mmHg or >21mmHg at the time of screening, or a difference in IOP between both eyes ≥5mmHg, or a previous diagnosis of ocular hypertension or glaucoma, or currently receiving any type of topical IOP-lowering (glaucoma) medication.
10. Received surgical intervention (ocular or systemic) within 6 months prior to the screening period, or planning to receive surgical intervention during the study period.
11. Use of any prohibited medication or treatment (ocular or periocular topical medication, systemic medication, injectable medication, and use of any lenses that can slow the progression of myopia) during the specified period before Visit 1. These medications or treatments are also prohibited during the study period. The shortest reasonable washout period for prohibited medications or treatments is:

    1. Any prescription or over-the-counter ophthalmic product (3 days); artificial tears are allowed, but not within 2 hours after the administration of the study drug.
    2. Monoamine oxidase inhibitors (7 days).
    3. Atropine, pirenzepine, or other anticholinergic drugs (60 days).
    4. Any medication affecting the pupil or accommodation (60 days).
    5. Orthokeratology (OK) lenses, rigid gas-permeable contact lenses, bifocal contact lenses, progressive multifocal lenses, multifocal contact lenses, or other lenses that can slow the progression of myopia (90 days).
    6. Monocular glasses and/or monofocal hydrophilic soft contact lenses for myopia correction can be normally used during the study period.
12. Expected use of ocular or systemic oral corticosteroids during the study period.
13. Participation in any other experimental treatment study within 30 days before the screening period or during the study period.
14. History or current disease that makes the subject prone to secondary myopia (e.g., Marfan syndrome, Stickler syndrome) or may affect visual function or development (e.g., diabetes, chromosomal abnormalities).
15. Presence of any condition or situation that the investigator believes may increase the risk to the subject, confound study data, or severely interfere with the subject's participation in the study, including but not limited to unstable: cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immune, skin, hematological, neurological, or psychiatric diseases.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2023-06-25 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Change in initial NITM (Nearwork-induced transient myopia) values from baseline to week 12. | DAY 1 & Week 12
  Compare the autorefractor NITM results measured in week 12 of the experimental and control group.

SECONDARY OUTCOMES:
Change from baseline in initial NITM values at week 2 and week 24 | Week 2 and week 24
  Measure the initial NITM (Near-Induced Transient Myopia) values at the designed time point.
Initial NITM values | Week 2
  Test the initial NITM (Near-Induced Transient Myopia) at each time point.
Initial NITM values | Week 12
  Test the initial NITM (Near-Induced Transient Myopia) at each time point.
Initial NITM values | Week 24
  Test the initial NITM (Near-Induced Transient Myopia) at each time point.
The difference between the change in initial NITM values | Day 1 & Week 12 & Week 24
  The difference between the change in initial NITM values from baseline to week 12 and the change from baseline to week 24

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoling Wang, Principal Investigator — Beijing Children's Hospital; Li Li, Principal Investigator — Beijing Children's Hospital
Locations (1):
- Beijing Children's Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No